CLINICAL TRIAL: NCT04004468
Title: Impact of Strength and Power Training on Golf Performance and Swing Biomechanics
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has left the institution.
Sponsor: Methodist University, North Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Project 2018 - 19 0027
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2019-08

CONDITIONS: Resistance Training With Traditional Periodization Model; Resistance Training With Conjugate Training Model
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Parallel groups participating in differing resistance training designs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Periodization Training (Active Comparator): Utilization of traditional periodization strength training model
  Interventions: Behavioral: Resistance Training
- Conjugate Training (Active Comparator): Utilization of conjugate strength model
  Interventions: Behavioral: Resistance Training

INTERVENTIONS:
Behavioral: Resistance Training — Standard barbell resistance training programs

SUMMARY:
Assess the impact of 10 weeks of strength and power training on Golf performance and swing biomechanics as measured by Trackman radar device and 16-camera monitoring system.

DETAILED DESCRIPTION:
Golf-specific exercise programs have been shown to improve strength, flexibility, and balance in golfers (1) and golf-specific plyometric training programs have been shown to significantly improve club head speed and ball carry distance in skilled adolescent golfers (2). Further, leg power, upper body strength, and arm strength have positively correlated with golf performance measures; most notably measures of distance and total score (3). The purpose of this study is to assess the effect of a 10-week strength and power training program on the biomechanics of the golf swing and golf performance.

Participants will have anthropometric data taken, including height, weight, and body composition.

Golf swing biomechanics will be assessed utilizing high-speed motion analysis cameras and software available in the Motion Analysis Laboratory in the McLean Health Sciences Building. The participant will don garments that fit snug to the skin and light-sensitive reflective markers will be placed on the subject. The motion of the swing will be captured utilizing the 14 camera Vicon Bonita 10 system with the Motion Monitor real-time Vicon plug-in. Club head speed will be assessed utilizing a Tracman 4 dual radar tracking system.

Power output for participants will be measured by performing a countermovement vertical jump and a static vertical jump on the 4 Bertec non-conductive forceplate system.

Strength assessments will be performed in the Nimocks Fitness Center by the Lead Investigator. Maximal strength will be assessed in the following lifts utilizing the parameters described by the National Strength and Conditioning Association (4): Back Squat; Flat Bench Press. Other maximal strength numbers for primary lifts involved in the program (Front Squat; Incline Bench; Power Cleans) will be prescribed as percentages of the tested lifts as follows: Maximal Front Squat = 80% of Maximal Back Squat; Maximal Incline Bench = 80% of Maximal Flat Bench; Maximal Power Clean = 70% of Maximal Back Squat.

ELIGIBILITY:
Inclusion Criteria: college aged golfers with no contraindications to exercise as measured by PAR-Q+

* No history of Heart condition or uncontrolled hypertension
* No history of chest pain at rest or with exertion
* No history of loss of balance or dizziness at rest or with exercise in previous 12 months
* No medications for chronic medical conditions
* No bone, joint, or soft tissue issue that could be made worse by becoming more physically active

Exclusion Criteria: As indicated by PAR-Q+

* History of arthritis, osteoporosis, or chronic back issues
* Current, or recent history of, cancer
* Diagnosed cardiovascular disease: CAD, heart failure, diagnosed abnormality of heart rhythm
* Uncontrolled high blood pressure (resting blood pressure of 160/90 or greater)
* Diagnosed Metabolic Condition: Type 1 diabetes, Type 2 diabetes, Pre-diabetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-05-05 (Estimated); Study Completion 2020-05-05 (Estimated)

PRIMARY OUTCOMES:
Gold club head speed and radar predicted 5-iron distance | 12 weeks
  Trackman measured club head speed and predicted carry of 5 iron
Biomechanics of golf swing | 12 weeks
  Bonita 16 camera measured biomechanical swing analysis

CONTACTS AND LOCATIONS:
Overall Officials: Blake Justice, Principal Investigator — Methodist University
Locations (1):
- Methodist University, Fayetteville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No